CLINICAL TRIAL: NCT04517773
Title: "Patient Autonomie" in People With Cancer
Acronym: AUPAC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: University of Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: AUPAC-IPC 2020-008
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Psychological; Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: Oncological patients
  Interventions: Other: writting test

INTERVENTIONS:
Other: writting test — Patients will be invitated to fill a questionary about self-autonomy

SUMMARY:
In France, the notion of autonomy concerning the patient's place in the healthcare system has been written into legal texts for several years. This notion is also fully recognized in our society and in the medical field by caregivers. However, the notion of autonomy is polysemous and complex. There is no unambiguous definition given the existence of plural conceptions of autonomy, especially in the field of psychology. A precedent thesis on the "representation of the autonomous patient in decision-making in the context of recurrence". Physicians practicing in oncology have been asked to perform a verbal association task inviting them to evoke the 5 words or expressions that came to their mind following the inductive word "autonomous patient". The results shows that for doctors, the "autonomous patient" is a patient with all of his physical, motor and intellectual capacities. Based on these findings, it would be interesting to study the autonomy perceived by the patient himself.

DETAILED DESCRIPTION:
In France, the notion of autonomy concerning the patient's place in the healthcare system has been written into legal texts for several years (Loi Kouchner, 2002; Loi Leonetti, 2005; Loi Leonetti-Claeys, 2016, etc.) . In addition,government policies are trying to adapt a strategy for transforming the health system. One of the priorities is to place "the patient at the heart of the system ". This orientation of positioning the patient at the center of the healthcare system taken by the Government, proves the importance of a contemporary reflection on the subject of the patient's autonomy. This notion is also fully recognized in our society and in the medical field by caregivers. Indeed, it constitutes a fundamental right of respect for the patient to decide for himself - in particular at the level of his health - what seems to be suitable, his therapeutic plan, his care, etc. However, the notion of autonomy is polysemous and complex. There is no unambiguous definition given the existence of plural conceptions of autonomy, especially in the field of psychology. Thus, through the literature, it can be understood as a psychological state, a personality variable, an attitude, a value, even a standard (Auzoult, 2008).

Given its omnipresence in public health, legislative, ethical, institutional as well as among caregivers, the investigators assume in our study that autonomy could be the object of social valuation and thus be understood as a shared norm. and conveyed. (Dubois & Beauvois, 2002). Norms are defined in particular as "cultural rules which guide behavior in a society" (Ross, 1973). In this perspective, the investigators can rely on the results of the work of Sonia Hadj Cherif's thesis on the "representation of the autonomous patient in decision-making in the context of recurrence". In this questionnaire survey of physicians practicing in oncology, the participants were asked to perform a verbal association task inviting them to evoke the 5 words or expressions that came to their mind following the inductive word "autonomous patient". The most salient elements associated with autonomy were: a good general state, management of daily life, valid, capacity for comprehension, hygiene, cognitive capacities preserved, movement, etc., thus representing the "autonomous patient" as a patient with all of his physical, motor and intellectual capacities. It is thus a functional autonomy in which the recognition of the patient depends first of all on his capacity to act and to do, which seems to prevail in medical discourse. Based on these findings, it would be interesting to study the autonomy perceived by the patient himself.

To do this, in our research, we will build a questionnaire intended for patients, the first part of which will be composed of a series of questions relating to the most significant associated words and their associated values for each patient to define his own representation of the "autonomous patient". The second part of the questionnaire will consist of three sub-questionnaires including items relating to patient autonomy. The items of these three questionnaires will be identical in all respects. Only the instruction requested from the patient will differ. In fact, patients will first of all be asked to respond as authentically as possible in order to situate their own perceived autonomy . Secondly, they will have to respond with a fictitious perspective of giving their doctor a favorable image of themselves. Finally, as a last step, they will have to give an unfavorable image of themselves to their doctor. These questionnaires will allow us to know whether cancer patients use different self-presentation strategies depending on whether they present to themselves, or to their doctor.

ELIGIBILITY:
Inclusion Criteria:

* All types of cancer;
* Minimum18 years old;
* Patients treated on the Paoli-Calmettes Institute;
* Non-objection of the patient following the information provided;
* Able to Read and understand;
* French Speaker;
* Affiliation to a social security scheme, or beneficiary of such a scheme.

Exclusion Criteria:

* cognitive disorders ;
* Patients at the end of their life.
* Person in an emergency situation, or unable to express a non-opposition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncological patients
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
words representing autonomy | day 0
  patient will write 5 words meaning autonomy for himself

SECONDARY OUTCOMES:
comparaition of "patients autonomy" for doctors and "patients autonomy" for patients | day 0

IPD SHARING:
Plan to Share IPD: No